CLINICAL TRIAL: NCT06282289
Title: Elicitation of Steady-state Audiovisual Responses in 6- and 10-month-old Infants
Acronym: AV-SSR-I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut de l'Audition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-077; 2023-A01798-37 (Other: ID RCB)
Record Dates: First submitted 2023-12-18; First posted 2024-02-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Speech
MeSH Terms: conditions — Speech | interventions — Magnetoencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-month-old infants (Other)
  Interventions: Behavioral: Magnetoencephalography (MEG); Other: Cognition development questionnaire
- 10-month-old infants (Other)
  Interventions: Behavioral: Magnetoencephalography (MEG); Other: Cognition development questionnaire

INTERVENTIONS:
Behavioral: Magnetoencephalography (MEG) — Stimuli will be presented binaurally through headphones at 60 decibel sound pressure level (dB SPL). Conditions are presented in a pseudo-random order with an inter-stimulus interval of ~800 ms on average (range: 600 ms to 1000 ms). The duration of the stimuli is fixed: 2 seconds, in order to guarantee a minimum number of cycles.
Other: Cognition development questionnaire — Computerised questionnaires completed by parents

SUMMARY:
The goal of this study is to investigate the preferential responses of speech neural systems in infants.

The main question it aims to answer is to determine whether the oscillatory synchronization capacity is associated with children's language level (i.e. vocabulary).

Participants will be presented with synthetically modulated stimuli at three frequency scales: 4 Hz, 5 Hz and 30 Hz.

ELIGIBILITY:
Inclusion Criteria:

* be 6 or 10 months old (+/- 2 weeks)
* have received age-appropriate information on the experiment
* their legal guardians have received appropriate information and given their oral consent.

Exclusion Criteria:

* A neurological disorder (visual, auditory, motor, executive)
* Developmental delay

Ages: 6 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
Significance of correlation between the delta (i.e. difference) of synchronization power estimated at 10- and 6-months of age and the delta of vocabulary level measured at 18months of age. | at 10-months, 6-months and 18-months of age

SECONDARY OUTCOMES:
The equation for linear regression analysis used to estimate the amount of neuronal synchronization between auditory and visual perception systems according to the Coherence and the Synchrony of AV inputs | at 10- and 6-months of age
The equation for linear regression analysis used to estimate the variation in the amount of neuronal synchronization between 4 experimental conditions according to the Coherence and the Synchrony of AV inputs | at 10- and 6-months of age
  4 experimental conditions : AV synchronous coherent, AV asynchronous coherent, AV synchronous incoherent, and AV asynchronous incoherent

IPD SHARING:
Plan to Share IPD: No